CLINICAL TRIAL: NCT00764998
Title: A Controlled Trial to Assess the Immunogenicity and Efficacy of Three Vaccine Dosing Strategies in HIV Infected Adults
Brief Title: Influenza Vaccine in HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario HIV Treatment Network (Network); Public Health Agency of Canada (PHAC) (Other Government); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CTN237
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Influenza; HIV
Keywords: Influenza; HIV; Influenza Vaccine; Efficacy
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Fluviral (Active Comparator)
  Interventions: Biological: Fluviral
- placebo (Placebo Comparator)
  Interventions: Biological: Fluviral

INTERVENTIONS:
Biological: Fluviral
  Other Names: non applicable

SUMMARY:
The purposes of this research study are:

1. to see if there is a difference in the quantity of protective influenza antibodies produced by different doses of the Fluviral vaccine
2. to see if these different vaccine dosing schedules reduce flu-like illness and/or reduce laboratory documented influenza in HIV Infected adults.

DETAILED DESCRIPTION:
Immune compromised individuals are at risk for infection with influenza and more likely to manifest more severe symptoms of influenza disease. Furthermore, they are influenza vaccine hyporesponsive in comparison to healthy, adult immune competent individuals. One population of immune compromised Canadians at risk for severe influenza disease is those living with HIV infection. At least 56,000 Canadians are HIV infected [1]. This population is at risk for more severe influenza illness. Influenza viral replication and shedding is prolonged and the duration of influenza symptomatology is longer in those with HIV [2, 3]. Furthermore, influenza-related mortality rates in HIV infected individuals are increased [4]. The HIV population is known to be hyporesponsive to vaccinations, including influenza. The efficacy of influenza vaccines is compromised, in part, by reduced antibody responses observed in HIV infected individuals [5]. Nevertheless, influenza vaccination is recommended for HIV-infected individuals [6, 7]. The Centers of Disease Control guidelines state: "Influenza can result in serious illness and because vaccination with inactivated influenza vaccine might result in the production of protective antibody titers, vaccination might benefit HIV-infected persons. Therefore, influenza vaccination is recommended". As influenza vaccination is the cornerstone of public health interventions intended to protect the population against influenza, vaccine hyporesponsiveness in immune compromised populations represents a significant concern. Given the risk of influenza exposure in general as well as concerns related to poor vaccine efficacy and more severe influenza disease in immune compromised populations such as those living with HIV, strategies to improve vaccine efficacy are required.

Therefore a total of 5 conditions provide justification for a trial to be conducted at this time:

1. current standard treatment with influenza vaccine is less efficacious when used in particular subgroups of immune compromised individuals, such as those diagnosed with HIV
2. there exists a significant burden of influenza infection in HIV patients that must be addressed in terms of identifying an effective treatment strategy
3. past randomized trials of influenza vaccination in HIV patients are of limited comparability to today's relevant base of patients, and alternative vaccination strategies require assessment
4. efficacy of booster doses of influenza vaccine in HIV patients remains in question as a consequence of methodologic shortcomings in terms of both design aspects and outcomes measured of past studies
5. there is a paucity of published evidence assessing the efficacy of an increased, double-dose of influenza vaccine in this patient population.

References

1. Boulos, D., et al., Estimates of HIV prevalence and incidence in Canada, 2005. Can Commun Dis Rep, 2006. 32(15): p. 165-74.
2. Safrin, S., J.D. Rush, and J. Mills, Influenza in patients with human immunodeficiency virus infection. Chest, 1990. 98(1): p. 33-7.
3. Radwan, H.M., et al., Influenza in human immunodeficiency virus-infected patients during the 1997-1998 influenza season. Clin Infect Dis, 2000. 31(2): p. 604-6.
4. Zanetti, A.R., et al., Safety and immunogenicity of influenza vaccination in individuals infected with HIV. Vaccine, 2002. 20 Suppl 5: p. B29-32.
5. Malaspina, A., et al., Compromised B cell responses to influenza vaccination in HIV-infected individuals. J Infect Dis, 2005. 191(9): p. 1442-50.
6. Health Canada Progress towards Canadian target coverage rates in Influenza and Pneumococcal Immunications., in Available at: http://www.phac-aspc.gc.ca/publicat/ccdr-rmtc/01vol27/dr2710eb.htlm. Accessed 8 December 2006. 2006.
7. Prevention and Control of Influenza. Recommendations of the advisory committee on immunization practice, in Centers for Disease Control and Prevention. Morbidity and Morality Weekly Report. 2006. p. Vol 55/RR-10.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - < 60 years
* HIV positive
* Able to provide signed, informed consent.

Exclusion Criteria:

* Receipt or anticipated requirement of any blood product, vaccine, or immunoglobulin preparation within one month of study vaccine administration until completion of study.
* Immunosuppressive therapy including prednisone, immune modulators, subjects undergoing dialysis, autoimmune dysfunction (including rheumatoid arthritis, lupus erythematosus, multiple sclerosis)
* Alcohol consumption > 4 drinks per day (1 drink is equal to a 12-ounce can of beer, or a 5-ounce glass of wine or one cocktail with 1 1/2-ounces alcohol)
* History of cancer, with the exception of cutaneous cancers including Kaposi Sarcoma, basal cell carcinoma and non-invasive HPV-related malignancy
* Known or suspected hypersensitivity to any component of the study vaccines, including chicken eggs or egg products and thimerosol
* History of immediate hypersensitivity reaction and/or reaction resulting in neurological symptoms to a previous dose of any influenza vaccine
* Presentation with or any recent history (within 24 hours) of any febrile illness (> 38 C) or symptoms of significant local or systemic infection - such subjects will be deferred from enrollment at least until one week after the illness has resolved
* Any other condition which in the opinion of the Investigator might interfere with evaluation of the study objectives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 285 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Immunogenicity measured by haemagglutination inhibition (HI) | baseline, week 4, week 8 and week 20.

SECONDARY OUTCOMES:
Frequencies of laboratory confirmed influenza and Frequencies clinical/respiratory illness | event driven

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Cooper, MD, Principal Investigator — OHRI
Locations (13):
- Canada (13):
  - Southern Alberta Clinic, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - BC Center for Excellence in HIV/Aids, Vancouver, British Columbia
  - Downtown Immunodeficiency Clinic / UBC, Vancouver, British Columbia
  - QEII HSC, Victoria General Hospital Site, Halifax, Nova Scotia
  - McMaster University Medical Center, Hamilton, Ontario
  - Infectious Disease Care Program, London, Ontario
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - University of Ottawa Health Services, Toronto, Ontario
  - Sunnybrook Health Science Center, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - HIV Care Program - Windsor Regional Hospital, Windsor, Ontario
  - Immunodeficiency Service, Montreal Chest Institute, Montreal, Quebec

REFERENCES:
- [Result] Cooper C, Thorne A, Klein M, Conway B, Boivin G, Haase D, Shafran S, Zubyk W, Singer J, Halperin S, Walmsley S; CIHR Canadian HIV Trials Network Influenza Vaccine Research Group. Immunogenicity is not improved by increased antigen dose or booster dosing of seasonal influenza vaccine in a randomized trial of HIV infected adults. PLoS One. 2011 Mar 25;6(3):e17758. doi: 10.1371/journal.pone.0017758. PMID 21512577
- [Derived] Nosyk B, Sharif B, Sun H, Cooper C, Anis AH; CIHR Canadian HIV Trials Network Influenza Vaccine Research Group. The cost-effectiveness and value of information of three influenza vaccination dosing strategies for individuals with human immunodeficiency virus. PLoS One. 2011;6(12):e27059. doi: 10.1371/journal.pone.0027059. Epub 2011 Dec 6. PMID 22162988